CLINICAL TRIAL: NCT02773069
Title: The Church as a Bridge to Deliver Health Resources Via Telehealth to Alleviate Obesity and Chronic Disease Disparities in Rural African Americans of Mississippi
Brief Title: The Church as a Bridge to Deliver Health Resources Via Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Collaborators: Southeast Mississippi Rural Health Initiative (Unknown); MSU Extension- Stone County (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R15MD010213-01 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Diet, Food, and Nutrition; Church; Healthcare Disparities; Minority Health; Mobile Health; Telehealth; Community-based Participatory Research; Primary Health Care; Weight Loss Programs; Health Behavior
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss program (Experimental): Participants will attend a 12 session weight loss program accompanied by maintenance support delivered by a church. Program will include peer education, telenutrition counseling and mobile health feedback.
  Interventions: Behavioral: Church Bridge Project

INTERVENTIONS:
Behavioral: Church Bridge Project — Community-based participatory research combining efforts of academic researchers, church leaders, primary care providers and community stakeholders.

SUMMARY:
The proposed Church Bridge intervention project will provide an innovative, evidence-based and technology supported, health intervention model for Southern, African American, and rural populations who continue to be disparately burdened by obesity and associated co-morbidities (i.e., hypertension, diabetes, cardiovascular disease). By targeting young adults (21-50 years of age) with families, the project will contribute to the long-term reduction of preventable chronic disease and related health care costs for the public.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/=30
* Must have elementary aged child (5-11 years) in household

Exclusion Criteria:

* Any health condition where weight loss is contraindicated
* Complicated disease states (ie., advanced renal disease or heart failure)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in weight at six months | 6 months